CLINICAL TRIAL: NCT02421887
Title: Males, Antioxidants, and Infertility (MOXI) Trial
Brief Title: Males, Antioxidants, and Infertility Trial
Acronym: MOXI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of North Carolina (Other); Augusta University (Other); Penn State University (Other); University of California, San Francisco (Other); University of Oklahoma (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOXI
Record Dates: First submitted 2015-03-19; First posted 2015-04-21 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidant Supplement (Active Comparator): Tablet: Vitamin C, 500 mg; Vitamin D3, 1000 IU; Vitamin E, 400 IU; Folic Acid 1000 mcg; Zinc, 20 mg; Selenium 200 mcg; Lycopene, 10 mg; Capsule: Vitamin D3, 1000 IU, L-Carnitine, 1000 mg
  Interventions: Drug: Antioxidant Supplement
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Antioxidant Supplement — An antioxidant combination including Vitamin C, Vitamin E, folic acid, selenium, zinc, and L-carnitine
  Arms: Antioxidant Supplement
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of the Males, Antioxidants, and Infertility (MOXI) Trial is to examine whether treatment of infertile males with an antioxidant formulation improves male fertility. The central hypothesis is that treatment of infertile males with antioxidants will improve sperm structure and function, resulting in higher fertilization rates and improved embryo development, leading to higher pregnancy and live birth rates. Findings from this research will be significant in that they will likely lead to an effective, non-hormonal treatment modality for male infertility. An effective treatment for men would also reduce the treatment burden on the female partner, lower costs, and provide effective alternatives to couples with religious or ethical contraindications to ART (Assisted Reproductive Technology). If antioxidants do not improve pregnancy rates, but do improve sperm motility and DNA integrity, they could allow for couples with male factor infertility to use less intensive therapies such as intrauterine insemination. Male fertility specialists currently prescribe antioxidants based on the limited data supporting their use. A negative finding, lack of any benefit, would also alter current treatment of infertile males.

ELIGIBILITY:
Inclusion Criteria:Couple

* 12 or more months of infertility (primary or secondary)
* Heterosexual
* Cohabitating and able to have regular intercourse

Male:

* ≥ 18 years of age
* At least one abnormal semen parameter on a semen analysis within the past 6 months:

  * Sperm concentration ≤15 Million/ml
  * Total motility ≤40%
  * Normal morphology (Kruger) ≤4%
  * DNA fragmentation (SCSA, DNA fragmentation index) >25%

Female:

* ≥18 years of age and ≤40 years of age
* For women ≥ 35 years of age, evidence of normal ovarian reserve as assessed by menstrual cycle day 3 (+/-2 days) FSH ≤10 IU/L with estradiol ≤ 70 pg/mL, AMH ≥ 1.0 ng/mL, OR antral follicle count >10 within one year prior to study initiation.
* Evidence of at least one patent fallopian tube as determined by an hysterosalpingogram or laparoscopy showing at least one patent fallopian tube or a saline infusion sonogram showing spillage of contrast material
* Regular cycles defined as ≥25 days and ≤35 days in duration
* Evidence of ovulation including biphasic basal body temperatures, positive ovulation predictor kits, or progesterone level ≥3 ng/ml.

Exclusion Criteria:

* Couple:

  * Previous sterilization procedures (vasectomy, tubal ligation). The prior procedure may affect study outcomes.
  * Planning in vitro fertilization in the next 6 months

Male:

* Sperm concentration < 5 million/mL on screening semen analysis
* Current use of a medication or drug that would affect reproductive function or metabolism (see Appendix C for list)
* Current multivitamin or herb use (requires 1 month wash-out)
* Current serious medical illnesses, such as cancer, heart disease, or cirrhosis
* Current use of anticoagulants
* Untreated hypothyroidism
* Uncontrolled diabetes mellitus

Female:

* History of surgically or medically confirmed moderate or severe endometriosis
* Body mass index >35 kg/m2
* Currently pregnant
* History of polycystic ovarian syndrome
* Current serious medical illnesses, such as cancer, heart disease, or cirrhosis
* History of systemic chemotherapy or pelvic radiation
* Current use of a medication or drug that would affect reproductive function or metabolism

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, Study Director — Eunice Kennedy Shriver National Institue of Child Health and Human Development; Nanette Santoro, MD, Study Chair — University of Colorado, Denver; Anne Z Steiner, MD, Principal Investigator — University of North Carolina; Michael P Diamond, MD, Study Director — Augusta University; Richard S Legro, MD, Study Director — Penn State University; Marcelle Cedars, MD, Study Director — University of California, San Francisco; Karl R Hansen, MD, Study Director — University of Oklahoma; Christos Coutifaris, MD, Study Director — University of Pennsylvania; Heping Zhang, PhD, Study Director — Yale University
Locations (10):
- United States (10):
  - Keck School of Medicine of University of Southern California, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Sunnyvale, California
  - Augusta University, Augusta, Georgia
  - Wayne State University, Southfield, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center - Women's Institute, Charlotte, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers through the NICHD DASH system. It will be available 6 months after publication of the primary results.
Time Frame: Following publication of the primary publication and when the de-identified data have been put into a format that is acceptable for DASH submission.

REFERENCES:
- [Derived] Spitzer TL, Trussell JC, Coward RM, Hansen KR, Barnhart KT, Cedars MI, Diamond MP, Krawetz SA, Sun F, Zhang H, Santoro N, Steiner AZ. Biomarkers of Stress and Male Fertility. Reprod Sci. 2022 Apr;29(4):1262-1270. doi: 10.1007/s43032-022-00853-x. Epub 2022 Feb 1. PMID 35106743
- [Derived] Steiner AZ, Hansen KR, Barnhart KT, Cedars MI, Legro RS, Diamond MP, Krawetz SA, Usadi R, Baker VL, Coward RM, Huang H, Wild R, Masson P, Smith JF, Santoro N, Eisenberg E, Zhang H; Reproductive Medicine Network. The effect of antioxidants on male factor infertility: the Males, Antioxidants, and Infertility (MOXI) randomized clinical trial. Fertil Steril. 2020 Mar;113(3):552-560.e3. doi: 10.1016/j.fertnstert.2019.11.008. Epub 2020 Feb 25. PMID 32111479
- See also: Related Info — http://c2s2.yale.edu/rmn/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antioxidant Supplement | Placebo
Started | 85 | 86
Completed | 68 | 77
Not Completed | 17 | 9
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Physician Decision | 2 | 4
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antioxidant Supplement | Placebo | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.0 [30.0 to 38.0] | 34.0 [30.0 to 37.0] | 34.0 [30.0 to 37.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 85 | 86 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 72 | 78 | 150
  Unknown or Not Reported | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 63 | 69 | 132
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Live Birth Rate
Time Frame: up to 15 months
Measure: Number; unit: percentage of live births
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 85 | 86
percentage of live births | 15.3 | 22.1

2. Secondary Outcome: Pregnancy Rate
Time Frame: up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 85 | 86
Participants | 18 | 26

3. Secondary Outcome: Miscarriage Rate
Description: miscarriages per total number of pregnancies
Time Frame: up to 9 months
Population: Miscarriage rate is calculated per number of participants who became pregnant.
Measure: Number; unit: miscarriages
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 18 | 26
miscarriages | 4 | 5

4. Secondary Outcome: Time to Pregnancy
Description: Time to pregnancy will be the chronologic time from randomization to pregnancy detection in days, in which the pregnancy is defined as a human Chorionic Gonadotropin (hCG) value over 5 on 2 separate occasions.
Time Frame: up to 7 months
Population: Time to pregnancy is calculated only for subjects who obtained pregnancy during the trial.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 18 | 25
days | 103.5 (62.3) | 123.5 (59.9)

5. Secondary Outcome: Change in Total Motile Sperm Count
Description: Samples will be assessed using a standard semen analysis
Time Frame: baseline and 3 months
Population: Participants for which semen samples were analyzed at both Baseline and Month 3 visit are included in this outcome measure.
Measure: Median (Inter-Quartile Range); unit: million sperm per mL
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 82 | 82
million sperm per mL | -4.0 [-13.2 to 9.9] | 1.5 [-11.8 to 15.4]

6. Secondary Outcome: Change in Deoxyribonucleic Acid (DNA) Fragmentation Index (DFI)
Description: DFI is the ratio of damaged sperm to total sperm. It is measured using Sperm Chromatin Structure Analysis (SCSA) which was performed on 5000 sperm per sample.
Time Frame: Baseline and 3 months
Population: Participants for which semen samples were analyzed for DFI at both Baseline and Month 3 visit are included in this outcome measure.
Measure: Mean (Inter-Quartile Range); unit: percentage of damaged DNA to total DNA
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 73 | 74
percentage of damaged DNA to total DNA | 18.7 [14.3 to 28.3] | 21.1 [14.1 to 28.6]

7. Secondary Outcome: Change in Semen Total Motility
Description: Samples assessed using a standard semen analysis
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: percentage of sperm with any motility
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 82 | 82
percentage of sperm with any motility | -1.6 (16.0) | -1.1 (13.7)

8. Secondary Outcome: Change in Sperm Concentration
Description: Samples assessed using a standard semen analysis
Time Frame: baseline and 3 months
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: million sperm per mL
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 82 | 82
million sperm per mL | -4.0 [-12.0 to 5.7] | 2.4 [-9.0 to 15.5]

9. Secondary Outcome: Change in Normal Morphology of Semen, Using World Health Organization (WHO) 5 Criteria
Description: Samples assessed using a standard semen analysis
Time Frame: baseline and 3 months
Population: Participants for whom semen samples were analyzed for morphology at both Baseline and Month 3 visit are included in this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percentage of sperm with normal morpholo
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 55 | 55
percentage of sperm with normal morpholo | 0 [-2.0 to 1.0] | 0 [-2.0 to 1.0]

10. Secondary Outcome: Change in Total Sperm Count
Description: Samples assessed using a standard semen analysis
Time Frame: baseline and 3 months
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: million sperm per sample
Arm/Group | Antioxidant Supplement | Placebo
Number analyzed (Participants) | 82 | 82
million sperm per sample | -10.6 [-32.5 to 12.6] | 1.6 [-21.8 to 42.9]

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from start of study drug through 30 days after the last dose of study medication, on average 7 months. Subjects completed a monthly diary where they reported any adverse events. They were also queried by study staff at each study visit about any adverse events since the last visit.
Arm/Group | Antioxidant Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/86
Other Adverse Events (participants affected / at risk) | 28/85 | 28/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antioxidant Supplement (N=85) | Placebo (N=86)
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Headache (General disorders) | 15 | 7
Nasopharyngitis (Infections and infestations) | 4 | 7
Nausea (Gastrointestinal disorders) | 1 | 4
Upper Respiratory Infection (Infections and infestations) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT02421887/Prot_SAP_ICF_000.pdf